CLINICAL TRIAL: NCT01477177
Title: Pilot Study of Polar Wand Carbon Dioxide Cryotherapy for Barrett's Esophagus With Low Grade and High Grade Dysplasia
Brief Title: Polar Wand Carbon Dioxide Cryotherapy for Barrett's Esophagus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment much slower than anticipated, and, funding issues
Sponsor: Mayo Clinic (Other)
Collaborators: Chek-Med Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Herbert C. Wolfsen, Professor of Medicine, Mayo College of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-004237
Record Dates: First submitted 2011-10-24; First posted 2011-11-22 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's esophagus dysplasia
MeSH Terms: conditions — Barrett Esophagus

ARMS (1):
- Polar Wand Treatment (Experimental): Cryotherapy device utilizing carbon dioxide (room temperature gas) for treatment of GI neoplasia
  Interventions: Device: Polar Wand carbon dioxide cryotherapy

INTERVENTIONS:
Device: Polar Wand carbon dioxide cryotherapy — Patients with Barrett's esophagus dysplasia will be treated with the Polar Wand device at 0 month, 2 and 4 months,6 months (with four quadrant surveillance biopsies), 8 and 10 months (treatment as necessary), and, at 12 months for final surveillance with biopsies throughout entire initial Barrett's segment length.

SUMMARY:
The purpose of this pilot study is to provide an initial assessment of the feasibility, safety and efficacy of Polar Wand carbon dioxide cryotherapy for treatment of Barrett's low grade and high grade dysplasia by use in a small number of patients so as to support, or otherwise, the development of a full-scale trial.

DETAILED DESCRIPTION:
Prospective pilot study to be performed in 14 Barrett's Esophagus patients with low grade and high grade dysplasia, referred for standard of care treatment. Patients will receive treatments with carbon dioxide Polar Wand cryotherapy at 0, 2 and 4 months, followed by surveillance endoscopy with four quadrant biopsies throughout the entire Barrett's esophagus (BE)segment at 6 months, followed by endoscopy with additional treatments (if needed) at 8 and 10 months, followed by a final surveillance endoscopy at 12 months, with four quadrant biopsies throughout the entire initial BE segment length.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for treatment with Barrett's esophagus with dysplasia as the original indication for ablative treatment.
* Previous fundoplication surgery is permitted
* Age 18 years to 98 years
* Ability to provide written, informed consent

Exclusion Criteria:

* Inability to obtain biopsies due to anticoagulation, varices, etc.
* Previous ablation therapy, wide area mucosal resection or external beam radiation to the thorax.
* Intolerance to twice daily proton pump inhibitor medication or inability to undergo sedation or endoscopic procedures.
* Worse than Grade B erosive esophagitis
* Less than 3 weeks from previous endoscopy with biopsy or 6 weeks from previous endoscopic therapy (resection).

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polar Wand Treatment
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Polar Wand Treatment
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 66 [61 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Barrett's Histology Grade, Using the Modified Vienna Classification
Description: The reduction of Barrett's segment length and histology classification will be measured at 12 months.
Time Frame: 12 months
Population: Terminated study. Enrollment much slower than anticipated and funding issues.
Arm/Group | Polar Wand Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Reduction in Barrett's Segment Length, Using the Prague Classification
Time Frame: 6 and 12 months
Population: Terminated study. Enrollment much slower than anticipated and funding issues.
Arm/Group | Polar Wand Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Assessment of Complications
Description: Specific complications are GI Bleeding and Perforation and Stricture and Ulceration
Time Frame: 12 months
Population: Terminated Study. Enrollment much slower than anticipated and funding issues
Arm/Group | Polar Wand Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Assessment of Post-ablation Symptoms
Description: Specific symptoms (frequency and severity) are chest pain, difficulty swallowing, painful swallowing, nausea or vomiting, sore throat
Time Frame: 12 months
Population: Terminated Study. Enrollment much slower than anticipated and funding issues.
Arm/Group | Polar Wand Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Reduction in Barrett's Histology Grade, Using the Modified Vienna Classification
Description: The reduction of Barrett's segment length and histology classification will be measured at 6 months.
Time Frame: 6 months
Population: Terminated Study. Enrollment much slower than anticipated and funding issues.
Arm/Group | Polar Wand Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for 12 months
Arm/Group | Polar Wand Treatment
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes